CLINICAL TRIAL: NCT00720447
Title: Phase II Study of Low Intensity Allogeneic Transplantation in Mantle Cell Lymphoma
Brief Title: Donor Stem Cell Transplant in Treating Patients With Mantle Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: UCL-BRD-07-137; CDR0000597903 (Registry Identifier: PDQ (Physician Data Query)); EUDRACT 2007-003081-18
Record Dates: First submitted 2008-07-19; First posted 2008-07-22 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2011-07

CONDITIONS: Lymphoma
Keywords: stage III mantle cell lymphoma; stage IV mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell | interventions — Alemtuzumab; Carmustine; Cytarabine; Etoposide; Melphalan; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: alemtuzumab
Biological: donor lymphocytes
Drug: carmustine
Drug: cytarabine
Drug: etoposide
Drug: melphalan
Procedure: allogeneic bone marrow transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Giving chemotherapy and monoclonal antibody therapy before a donor stem cell transplant helps stop the growth of cancer cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets.

PURPOSE: This phase II trial is studying donor stem cell transplant in treating patients with mantle cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine progression-free survival in patients with mantle cell lymphoma undergoing low-intensity allogeneic stem cell transplantation.

Secondary

* Determine overall survival of these patients.
* Determine the toxicity by way of adverse event profile of this regimen in these patients.

OUTLINE: This is a multicenter study.

* Reduced intensity conditioning: Patients receive carmustine IV over 2 hours on day -6, etoposide IV over 1 hour and cytarabine IV over 15 minutes on days -5 to -2, alemtuzumab IV over 2 hours on days -5 to -1, and melphalan IV on day -1.
* Donor stem cell transplant: Patients undergo stem cell transplantation on day 0 with filgrastim (G-CSF)-mobilized peripheral blood stem cells or bone marrow stem cells.
* Graft-versus-host disease (GVHD) prophylaxis: Patients receive cyclosporine IV or orally on day -1 to 30 and taper to day 100.
* Donor lymphocyte infusion (DLI) therapy: Patients with evidence of disease progression, mixed chimerism, or low level residual disease undergo DLI every 3 months for up to 15 months in the absence of GVHD.

After completion of study, patients are followed every 3 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of mantle cell lymphoma
* No relapsed or progressive disease
* Achieved at least a partial remission following induction chemotherapy
* HLA-matched donor available
* Blood samples from both patient and donor available for chimerism studies
* No central nervous system involvement

PATIENT CHARACTERISTICS:

* ECOG performance status 2-4
* Considered fit for transplant by treating physician
* Serum bilirubin ≤ 1.5 times upper limit of normal
* Alkaline phosphatase ≤ 2 times normal
* Creatinine clearance ≥ 50 mL/min
* Ejection fraction > 50% (no inadequate cardiac function)
* Not pregnant or nursing
* Negative pregnancy test
* No symptomatic respiratory compromise
* No serious concurrent disease which would preclude allograft
* No known serological positivity for hepatitis B, hepatitis C, or HIV
* No history of a psychological illness or condition that would affect compliance
* No previous malignancy within the past 5 years except nonmelanoma skin tumors or stage 0 (in situ) cervical carcinoma

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Overall survival
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Simon Rule, MD, Principal Investigator — Derriford Hospital